CLINICAL TRIAL: NCT05852379
Title: Transcutaneous Auricular Vagus Nerve Stimulation Paired With Rehabilitation and Pelvic Nerves Stimulation for Improvement Motor Functions of Lower Extremities in Peoples With Chronic Spinal Cord Injury
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Spinal Cord Injury
Acronym: taVNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Possover International Medical Center AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Possover International Medical
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Nervous System Diseases; Trauma, Nervous System; Movement Disorders; Central Nervous System Diseases
Keywords: gait; Vagus Nerve Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Nervous System Diseases; Trauma, Nervous System; Movement Disorders; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, parallel assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (participants, Care provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcutaneous auricular vagus nerve stimulation (Experimental): PtaVNS, twice daily, 30 minutes each time over 6 months. Followed by 6 months home excercice program, physiotherapy twice a week, and continuous low frequency antidromic pelvic neuromodulation (CAPN).
  Interventions: Device: active taVNS
- Sham transcutaneous auricular vagus nerve stimulation (Sham Comparator): Sham PtaVNS (fictive stimulation), twice daily, 30 minutes each time over 6 months. Followed by 6 months home excercice program, physiotherapy twice a week, and continuous low frequency antidromic pelvic neuromodulation (CAPN).
  Interventions: Device: sham taVNS

INTERVENTIONS:
Device: active taVNS — Transcutaneous auricular vague nerve stimulation
  Arms: Active transcutaneous auricular vagus nerve stimulation
Device: sham taVNS — Scham transcutaneous auricular vague nerve stimulation
  Arms: Sham transcutaneous auricular vagus nerve stimulation

SUMMARY:
This study is a single blinded prospective randomized monocentric study examining the effectiveness of transcutaneous auricular vagus nerve stimulation paired with rehabilitation and low frequency/antidromic stimulation of the pelvic somatic nerves. The investigator hypothesize that treatment using transcutaneous auricular vagus nerve stimulation will improve gait recovery in spinal cord injured participants already treating by rehabilitation and pelvic nerves neuromodulation.

DETAILED DESCRIPTION:
In this single-blinded prospective randomized study, 10 participants (adults above 18years) with chronic spinal cord injury already managed with active rehabilitation and continuous pelvic nerves stimulation (low-frequency, antidormic) will be randomly assigned in a 1:1 ratio to active taVNS (twice daily, 30 minutes each time), or control with daily sessions of sham taVNS (0.0 mA). Rehabilitation is performed unspecifically by home-rehabilitation's team or physiotherapeutists with exercises adjusted to the participant's functional level. This protocol comprised 15 to 20 weekly hours of multidisciplinary care, including neurofunctional physiotherapy and aquatic therapy, cardiorespiratory physiotherapy (two hours/week). All participants have undergone previously an implantation of a stimulator for chronic neuromodulation of the pelvic somatic nerves according with the LION procedure. Participants and therapeutists will maintain blinding until the completion of the study (6 months). Assessment of gait function, motor symptoms are performed three time, at baseline, at 3-months follow up and at 6months follow up.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of traumatic complete/incomplete apar/teraplgia
* At least 12 months post-traumatic SCI
* Patient included in rehabilitation program
* After laparoscopic implantation of neurosprothesis to the pelvic nerves (LION procedure)
* Mini-mental State examination score>24
* Stable medication
* Patient who voluntarily accept the test and sign an informed consent form

Exclusion Criteria:

* There is a clear history of cerebrovascular stroke, and there are clear symptoms or signs of neurological deficit at the time of onset, and there are corresponding responsible lesions left on neuroimaging
* Patients with significant visual impairment or coexisting local or systemic diseases (eg osteoarthritis, or neuro,ogical conditions) likely to affect gait are excluded from the study
* Pathologies of the articulation and ligaments of the LE that make standing/walking anatomically impossible
* Patients who underwent deep brain stimulation surgery or those with an implanted cardiac pacemaker are excluded
* Those with history of alcoholism, or drug addiction, or neurological diseases that can cause cognitive impairment, such as brain injury, epilepsy, encephalitis, normal intracranial pressure hydrocephalus
* Suffering from systemic diseases that may lead to cognitive impairment (such as liver and kidney insufficiency, endocrine diseases, vitamin deficiency)
* Suffering from cardiac conductive dysfunctions or sleep apnea syndrome
* Participating in other drug clinical trials
* There are contraindications to head MRI
* Those who are deemed unsuitable to participate the trial by the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the Walking Index for Spinal Cord Injury (WISCI II | 6 months
  Standardized scale that classifies the individual's walking ability in 21 levels,from 0 to 20 (Table 2), from the preoperative to the 6-month assessment. (Morganti B, Scivoletto G, Ditunno P, Ditunno JF, Molinari M. Walking index for spinal cord injury (WISCI): criterion validation. Spinal Cord 2005;43:43-71)

SECONDARY OUTCOMES:
ASIA Lower Extremity Motor | 6 months
  Motor Scoring (scoring on reverse side) L2: Hip flexors L3: Knee extensors L4: Ankle dorsiflexors L5: long toe extensors S1: ankle platter flexors
  Scores:
  0: total paralysis
  1. palpable or visible contraction
  2. active movement, gravity eliminated
  3. active movement, against gravity
  4. active movement; against some resistance
  5. active movement, against full resistance

CONTACTS AND LOCATIONS:
Overall Officials: Marc MP Possover, MD, PhD, Principal Investigator — Possover International Medical Center AG - Klausstrasse 4, CH-8002 Zürich

IPD SHARING:
Plan to Share IPD: No